CLINICAL TRIAL: NCT04972448
Title: A Clinical Translational Study on the Multi-gene Assays and RecurIndex for Predicting the Breast Cancer Recurrence Risk in Cross-strait Chinese Patients With Early-stage Luminal Breast Cancer
Brief Title: RecurIndex Predicts Risk of Recurrence in Early-stage Luminal Breast Cancer
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: ZhejiangCH-0709
Record Dates: First submitted 2021-07-12; First posted 2021-07-22 (Actual); Last update posted 2021-07-22 (Actual); Status verified 2021-07

CONDITIONS: Breast Cancer; Recurrence
MeSH Terms: conditions — Breast Neoplasms; Recurrence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Group1: Chemotherapy+endocrine therapy+radiotherapy
- Group2: Chemotherapy+endocrine therapy
- Group3: endocrine therapy+radiotherapy
- Group4: endocrine therapy

SUMMARY:
This study will conduct a multicenter, open, prospective clinical trial to observe the RecurIndex to assist in predicting the risk of recurrence in patients with early-stage Luminal-type breast cancer. The aim of this study is to validate the predictive effect of the RecurIndex on the risk of recurrence in women with early-stage Luminal-type breast cancer in China.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old, ≤ 70 years old.
* Eastern Cooperative Oncology Group (ECOG) ≤ 2.
* Postoperative pathology is clearly diagnosed as invasive breast cancer.
* Estrogen receptor (ER) or progesterone receptor (PR) positive, HER2 negative.
* Available with Formalin-Fixed and Parrffin-Embedded (FFPE) tumor tissue.
* Stage I-II patients who have received surgery (breast-conserving or mastectomy) and the pathological staging is pT1-2N0-1M0 or pT3N0M0.
* The patient had not received systemic systemic treatment (including radiotherapy, chemotherapy, immunotherapy, endocrine therapy) before enrollment.
* Signed an informed consent form.

Exclusion Criteria:

* Breast cancer patients whose clinical or pathological stage is T4, N2-3 or M1.
* Known human immunodeficiency virus infection (HIV) or acquired immunodeficiency syndrome (AIDS) related diseases.
* Other psychiatric disorders that may interfere with the judgment of the study results, or abnormal laboratory tests; and who, in the judgment of the investigator, are considered unfit to participate in the study.
* Patients with double breast cancer.
* Severe/uncontrolled intercurrent diseases/infections.
* Subjects with allogeneic organ transplants requiring immunosuppressive therapy.
* Hormone receptors ER and PR are negative (any detectable estrogen and progesterone receptors do not express or express <1%) and/or HER2 overexpression/amplified by FISH detection.
* Not suitable for hormone receptor modulators (e.g. tamoxifen) and adjuvant endocrine other drug therapy.

Ages: 18 Years to 70 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Women with breast cancer
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2021-07 (Estimated); Primary Completion 2025-05 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
invasive disease-free survival (IDFS) | 5 years
  defined as time between treatment and the time of invasive disease occurred
recurrence free survival (RFS) | 5 years
  defined as time between treatment and the time of any recurrence of ipsilateral chest, breast, regional lymph node recurrence, distant metastases, or death occurred

SECONDARY OUTCOMES:
overall survival (OS) | 5 years
  defined as time between treatment and the time of death occurred
distance metastasis-free interval (DMFI) | 5 years
  defined as time between treatment and the time of distant metastases, or death
local-regional recurrence-free interval (LRFI) | 5 years
  defined as time between treatment and the time of any recurrence of ipsilateral chest, breast, regional lymph node recurrence, distant metastases, or death occurred

CONTACTS AND LOCATIONS:
Overall Officials: Xiajia Wang, MD, Study Chair — Zhejiang Cancer Hospital